CLINICAL TRIAL: NCT04020328
Title: A Randomized, Controlled Trial to Evaluate Leflunomide Plus Low Dose Corticosteroid Therapy in Progressive IgA Nephropathy With Renal Insufficiency
Brief Title: Leflunomide Plus Low Dose Corticosteroid in Immunoglobulin A (IgA) Nephropathy With Renal Insufficiency
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, XUYI, Principal Investigator, Shenzhen Second People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20193357002
Record Dates: First submitted 2019-07-10; First posted 2019-07-16 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Glomerulonephritis, IGA; Renal Insufficiency, Chronic
Keywords: Leflunomide; Glucocorticoids; Conservative Treatment; Glomerulonephritis, IGA; Renal Insufficiency, Chronic
MeSH Terms: conditions — Glomerulonephritis, IGA; Renal Insufficiency, Chronic | interventions — Leflunomide; Prednisone

STUDY DESIGN:
Intervention Model Description: the participants who met the inclusion and exclusion criteria were randomly assigned to leflunomide + low dose glucocorticoids treatment group and conservative treatment group in a 1:1 ratio
Masking Description: it is a open label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- leflunomide + low dose glucocorticoids therapy group (Experimental): the experimental group will receive leflunomide + low dose glucocorticoids therapy on the basis of conservative treatment, while the control group receive conservative treatment
  Interventions: Drug: Leflunomide 20 mg+prednisone 0.5mg/kg/d
- Basic conservative treatment group (No Intervention): the basic conservative treatment group is the delaying the progress of renal function, including low-protein diet supplemented with ketoacid therapy, RAS inhibitor, blood pressure control, lipid-regulating therapy and antiplatelet aggregation therapy

INTERVENTIONS:
Drug: Leflunomide 20 mg+prednisone 0.5mg/kg/d — Leflunomide plus low dose glucocorticoids to have the immunosuppressive therapy to those progressive IgA nephropathy with eGFR<50ml/min
  Other Names: Arava
  Arms: leflunomide + low dose glucocorticoids therapy group

SUMMARY:
IgA nephropathy is the most common primary glomerulonephritis in the world. Because of the poor treatment effect in advanced patients, it is still the main cause of maintenance dialysis. Current immunosuppressive therapy is still controversial, especially to those progressive IgA nephropathy with eGFR<50ml/min. Leflunomide is widely used in the treatment of rheumatic diseases, such as rheumatoid arthritis and lupus nephritis, it's serum concentration will not be affected by renal function, and it also has antiviral effect. There are two randomized controlled trials and a retrospective study suggesting that leflunomide combined with glucocorticoids can effectively control urinary protein compared with glucocorticoids or conservative treatment, but these three studies are not specifically targeted at patients with estimated Glomerular Filtration Rate(eGFR) < 50ml/min.

Investigators will perform a prospective, open-label, randomized, controlled trial to evaluate the efficacy and safety of leflunomide and low dose glucocorticoids therapy in progressive IgA nephropathy with eGFR<50ml/min

DETAILED DESCRIPTION:
all the participants enrolled in the study will be randomly assigned in a 1:1 ratio, the experimental group will receive leflunomide + low dose glucocorticoids therapy on the basis of conservative treatment, while the control group receive conservative treatment only. Conservative treatment is defined as the treatment of delaying the progress of renal function, including low-protein diet supplemented with ketoacid therapy, Renin Angiotensin system (RAS) inhibitor, blood pressure control, lipid-regulating therapy and antiplatelet aggregation therapy. The course of treatment will last one year, then the leflunomide+glucocorticoids group will continue the conservative treatment. Participants will be follow-up at least 98 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 14 to 65 years old participants, No restrictions on gender or race
* Diagnosis of primary IgA nephropathy
* Renal biopsy within 6 months before screening. Renal pathology shows diffuse IgA deposition in the Mesangial area and dense deposition in the Mesangial area under electron microscope. glomeruli more than 8
* persistent proteinuria ≥ 1 g/24 hr (or urine protein/creatinine ratio ≥ 1.0 mg/g), eGFR at 25-50 ml/min/1.73 m2 (calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula)
* signed written consent; patients under 18 years old need to have legal guardians to sign informed consent at the same time

Exclusion Criteria:

* Secondary IgA nephropathy (such as lupus nephritis, Henoch-Schönlein purpura, hepatitis B associated glomerulonephritis, hepatitis C associated glomerulonephritis, liver cirrhosis and other autoimmune diseases)
* eGFR < 25 ml/min/1.73m2 or eGFR > 50 ml/min/1.73m2 (calculated by CKD-EPI formula)
* Special types of IgA nephropathy need to be excluded, such as crescent IgA glomerulonephritis (defined as the presence of crescents in over 50% of the glomeruli), or minimal lesions with IgA deposition
* Acute kidney injury within 3 months before screening
* Received immunosuppressive therapy within 3 months before screening
* Patients who had acute or chronic infections that need treatment, and the researchers judged that they were not suitable for inclusion in the study
* Pregnancy, lactation or unreliable birth control
* Dialysis treatment before screening
* Allergic or taboo to planned drugs (such as leflunomide, glucocorticoids, etc.)
* Severe acute or chronic diseases that the researchers believe may bring an excessive risk to the subjects
* A history of malignant tumors within 5 years, with the exception of carcinoma in situ and papillary thyroid carcinoma which have been adequately treated
* Participated in other clinical trials and / or used other research drugs within 4 weeks prior to screening

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
renal survival rate | at least 96 weeks
  50% increase in serum creatinine compared with the baseline level or End Stage Renal Disease(ESRD)

SECONDARY OUTCOMES:
proteinuria | at least 96 weeks
  changes in proteinuria compared to the baseline
eGFR | at least 96 weeks
  extent of eGFR decline compared with the baseline and annual decline rate
complete remission rate | at least 96 weeks
  Complete Remission (CR): proteinuria < 1.0g / 24hr, Scr stable (Scr increase ≤ 15% baseline level)
partial remission rate | at least 96 weeks
  Partial Remission (PR): proteinuria in 1.0-3.5g/24hr range and decrease more than 50%, Scr stable (Scr increased ≤ 15% baseline level)
no response rate | at least 96 weeks
  No Response (NR)：proteinuria > 3.5g/24hr or decrease less than 50% of baseline , with or without deterioration of renal function

CONTACTS AND LOCATIONS:
Locations (1):
- Xu Yi, Shenzhen, Guangdong, China

REFERENCES:
- [Derived] Alladin A, Hahn D, Hodson EM, Ravani P, Pfister K, Quinn RR, Samuel SM. Immunosuppressive therapy for IgA nephropathy in children. Cochrane Database Syst Rev. 2024 Jun 12;6(6):CD015060. doi: 10.1002/14651858.CD015060.pub2. PMID 38864363